CLINICAL TRIAL: NCT04142684
Title: Phrenic Nerve Conduction Study to Diagnose Unilateral Diaphragmatic Paralysis
Acronym: ENMG-DIAPH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190618
Record Dates: First submitted 2019-09-26; First posted 2019-10-29 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: Unilateral Diaphragmatic Paralysis
Keywords: Unilateral Diaphragmatic Paralysis; Diagnose; Phrenic Nerve
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims as the principal objective to compare two approaches to diagnosis unilateral diaphragmatic paralysis: transdiaphragmatic pressure (Pdi) measurement versus phrenic nerve conduction (NPC) study.

The secondary objective of the study is the strengths and weaknesses of different tests. Diagnostic threshold values.

DETAILED DESCRIPTION:
Inpatient patients in Raymond Poincaré hospital are informed of the utilization of their data retrospectively by the hospital's welcome booklet and reports of patients' hospitalization.

Period of date collected: November 2015 to June 2018.

The reference standard was the diagnosis established during a multidisciplinary meeting held during patient management involving a neurologist, an electrophysiologist, a pulmonologist, and a respiratory physiologist. The medical history, physical findings, and all available investigations including imaging studies, ENMG, lung function tests, and Pdi measurement were considered during the meeting.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years;
* Available data of Pdi and PNC;
* Suspected unilateral diaphragmatic paralysis.

Exclusion Criteria:

* Abnormalities in thoracic wall which susceptible to modify the investigation's results;
* Scoliosis;
* Pleural effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suspected unilateral diaphragmatic paralysis with available Pdi and PNC data.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Diaphragm evaluation-compound muscle action potential | at 1 month
  Right and left diaphragm compound muscle action potential (CMAP) : CMAP of Right and left diaphragm were elicited by transcutaneous electrical stimulation of phrenic nerves at the posterior edge of the sternocleido mastoid muscle. They are recorded with two surface electrodes positioned in the eighth intercostal space. The intensity of electrical stimulation was increased until no additional increment in diaphragm CMAP was observed. CMAP amplitude of 300µV or greater and latencies of 9 milliseconds or less were considered normal.
Diaphragm evaluation-transdiaphragmatic pressure | at 1 month
  Transdiaphragmatic pressure (Pdi) was computed as the difference between gastric and esophageal pressure. Pdi was considered normal when magnetic stimulation of both phrenic nerves induced a Pdi change (Pdi Twitch) above 18 cmH2O and unilateral stimulation of each nerve induced a Pdi change (unilat-Pdi Twitch) above 4 cmH2O and ratio of the two unilat-Pdi Twitch > 0.5. and < 2.

SECONDARY OUTCOMES:
Spirometry | 1 month
  Spirometry will be performed in the upright and supine positions. Upright vital capacity (VC) was reported as % predicted value and the difference between upright and supine VC (VC) as % upright value (normal value > 75%).
Lung volume measurements | 1 month
  Lung volume measurements will be performed in the upright and supine positions. Upright vital capacity (VC) was reported as % predicted value and the difference between upright and supine VC (VC) as % upright value (normal value > 75%).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LOFASO, MD, PhD, Principal Investigator — Service de Physiologie et Explorations Fonctionnelles, Hôpital Raymond Poincaré, APHP, Garches, FRANCE; Vivien REYNAUD, MD, Study Director — Service de Physiologie et Explorations Fonctionnelles, Hôpital Raymond Poincaré, APHP, Garches, FRANCE
Locations (1):
- Service de Physiologie et Explorations Fonctionnelles, Hôpital Raymond Poincaré, APHP, France, Garches, France

IPD SHARING:
Plan to Share IPD: No